CLINICAL TRIAL: NCT06565520
Title: Modulating Cortical Excitability to Improve Functional Movements in Individuals With Patellofemoral Pain: a Randomized Control Trial
Brief Title: Modulating Cortical Excitability to Improve Functional Movements in Individuals With Patellofemoral Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UNLV-2022-69
Record Dates: First submitted 2024-08-07; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) (Experimental)
  Interventions: Device: transcranial direct current stimulator
- Sham (Sham Comparator)
  Interventions: Device: transcranial direct current stimulator

INTERVENTIONS:
Device: transcranial direct current stimulator — The total amount of participation time per qualified subject will be approximately 150 minutes over two sessions. The participant screening session will take approximately 30 minutes, which is an appropriate amount of time to complete all screening tasks. The tDCS and sham sessions will take approximately a total of 120 minutes over two sessions.
  The first session will include a screening (30 minutes) to ensure they qualify for the study, followed by a treatment session (60 minutes): including non-invasive brain stimulation combined with hip strengthening exercises and functional movement testing at UNLV Maryland Campus. Subjects will return for a second treatment session (60 minutes) 2 weeks after the first.

SUMMARY:
This study sought to investigate whether modulation of cortical excitability of the gluteal musculature, via tDCS paired with exercise, will reduce the amount the knee caves in during functional tasks in individuals with PFP. The objective is the explore if having tDCS target the area of the brain controlling hip muscles, when paired with exercise, will be more effective in reducing the amount the knee caves in for individuals with PFP versus those who receive exercise alone as their treatment. The aim is to contribute our findings to the growing knowledge in this area in order to help establish the possibility, and feasibility, of its use in clinical settings to strengthen traditional treatments for this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. are between 18 and 45 years old
2. have had patellofemoral pain (PFP; kneecap pain) on one side for at least 3 months, and 3) the knee does cave in when performing functional movements.

Exclusion Criteria:

1. do not have pain coming from the kneecap during screening;
2. have a history of knee injury or surgery,
3. have a history of seizures and/or taking anti-seizure medication,
4. have an implanted device that interacts with electric current,
5. have a history of balance disorder,
6. currently are pregnant or think they may be pregnant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-04-21 (Estimated); Study Completion 2025-04-21 (Estimated)

PRIMARY OUTCOMES:
trunk lean angle | Baseline and Immediately after intervention
knee frontal plane projection angle | Baseline and Immediately after intervention
hip frontal plane projection angle | Baseline and Immediately after intervention
dynamic valgus index | Baseline and Immediately after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kai Yu Ho, PhD, Principal Investigator — UNLV
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No